CLINICAL TRIAL: NCT00099294
Title: A Randomized Phase 3 Study of the Efficacy and Safety of Glufosfamide Compared With Best Supportive Care in Metastatic Pancreatic Adenocarcinoma Previously Treated With Gemcitabine
Brief Title: Study of the Efficacy and Safety of Glufosfamide Compared With Best Supportive Care in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-302
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Cancer; Pancreatic Adenocarcinoma; Metastatic; Glufosfamide
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — beta-D-glucosylisophosphoramide mustard

INTERVENTIONS:
Drug: Glufosfamide

SUMMARY:
The primary objectives of the study is to evaluate the effectiveness and safety of glufosfamide in subjects with pancreatic cancer who have been previously treated with gemcitabine as measured by overall survival compared with best supportive care.

DETAILED DESCRIPTION:
TH-CR-302 is a randomized Phase 3 study that will evaluate the efficacy and safety of glufosfamide plus best supportive care (BSC) compared to BSC alone for second line treatment of metastatic pancreatic cancer. BSC includes all medical or surgical interventions that a pancreatic cancer patient should receive to palliate the cancer but excludes treatment with systemic therapies intended to kill the cancer cells.

Study Hypothesis: Glufosfamide will provide benefits in survival to patients with metastatic pancreatic cancer over best supportive care.

Comparison: Glufosfamide versus best supportive care.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Pancreatic adenocarcinoma proven either by histology (surgical biopsy) or cytology (CT- or endoscopic-guided)
* Metastatic pancreatic cancer
* Disease progression during or after treatment with gemcitabine (alone or in combination with other agents; at regular, not radiosensitizing, doses) for advanced/metastatic pancreatic cancer
* Measurable or nonmeasurable disease by RECIST criteria (at least one target or nontarget lesion)
* Recovered from reversible toxicities of prior therapy
* Karnofsky performance status ≥70
* All women of childbearing potential and all men must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) from entry into the study through 6 months after the last dose
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee

Exclusion Criteria:

* More than one prior systemic therapy regimen for metastatic/locally advanced pancreatic cancer (radiosensitizing doses of 5FU or gemcitabine at the time of initial radiotherapy do not count as a prior systemic therapy regimen)
* Hormonal therapy, radiation therapy, biologic therapy, chemotherapy or other systemic antitumor therapy for pancreatic cancer within 14 days prior to study start
* Symptomatic brain metastases (baseline CT scan is not required in asymptomatic subjects)
* Active clinically significant infection requiring antibiotics
* Known HIV positive or active hepatitis B or C
* Recent (one year) history or symptoms of cardiovascular disease (NYHA Class 2, 3, or 4), particularly coronary artery disease, arrhythmias or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, or congestive heart failure
* No other active malignancies (other than treated non-melanoma skin cancer or treated in situ cancer) within the past year
* Major surgery within 3 weeks of the start of study treatment, without complete recovery
* Clinically significant abnormalities in laboratory test results (including complete blood count, chemistry panel including electrolytes, and urinalysis) (Hemoglobin <9 g/dL (may receive transfusion or erythropoietin to maintain))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival

SECONDARY OUTCOMES:
Objective tumor response rate
Duration of objective tumor response rate
Progression-free survival
6 month and 12 month survival
Serum CA 19-9
Pain Intensity
Performance Status

CONTACTS AND LOCATIONS:
Locations (111):
- United States (23):
  - Augusta Oncology Associates, Los Angeles, California
  - Kenmar Research Institute, Los Angeles, California
  - Mile High Oncology, Denver, Colorado
  - Northwestern Connecticut Oncology - Hematology Associates, Torrington, Connecticut
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - Hematology/Oncology of the North Shore, Skokie, Illinois
  - Fort Wayne Medical Oncology/Hem, Fort Wayne, Indiana
  - Norton Healthcare Center, Louisville, Kentucky
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Hattiesburg Clinic Oncology, Hattiesburg, Mississippi
  - Columbia Comprehensive Cancer Care Clinic, Columbia, Missouri
  - Bond Clinic, Rolla, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Office of Clinical Trials, Paramus, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Hanover Medical Specialists, Wilmington, North Carolina
  - Vita Hematology Oncology PC, Bethlehem, Pennsylvania
  - The Family Cancer Center , PLLC, Collierville, Tennessee
  - Center for Oncology Research and Treatment, Dallas, Texas
  - JPS Center for Cancer Care, Fort Worth, Texas
  - Northern Utah Associates, Ogden, Utah
  - Cancer Outreach Association, Abingdon, Virginia
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Argentina (8):
  - Hospital Interzonal General de Agudos, Buenos Aires
  - Hospital Posadas, Buenos Aires
  - Policlinica Privada Instituto de Medicina Nuclear, Buenos Aires
  - Hospital Udaondo, Buenos Aires
  - Hospital Alvarez, Buenos Aires
  - Hospital Churruca - Visca, Buenos Aires
  - Instituto Medico Alexander Fleming, Buenos Aires
  - Instituto CAICI, Santa Fe
- Brazil (11):
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Hospital Vera Cruz - Clinica de Oncologia, Belo Horizonte
  - Hospital Luxemburgo, Belo Horizonte
  - Hospital de Clínicas da UFPR, Curitiba
  - Associacao de Combate ao Cancer em Goias, Hospital Araujo Jorge, Setor de Oncologia Clinica, Goiânia
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - Instituto Nacional do Cancer - INCA, Rio de Janeiro
  - Grupo Paulista Oncologia Integrada, São Paulo
  - Clinica de Oncologia Medica S/C Ltda, São Paulo
  - Hospital do Cancer - AC Camargo, São Paulo
- Bulgaria (8):
  - Department of Chemotherapy Dr. Georgi Stranski General Hospital of Pleven University, Pleven
  - First Internal Department Plovdiv Regional Oncology Center with In-patient Department, Plovdiv
  - Department of Chemotherapy Sofia Regional Oncology Center, Sofia
  - Chemotherapy Clinic Queen Joanna General Hospital, Sofia
  - Haematology and Oncology Clinic Military Medical Academy, Sofia
  - Chemotherapy Clinic Specialized Oncology Hospital, Sofia
  - Department of Medicinal Oncotherapy and Palliative Care Dr. Marko Markov Regional Oncology Center, Varna
  - Department of Chemotherapy Veliko Tarnovo Regional Oncology Center, Veliko Tarnovo
- Czechia (5):
  - Fakultni nemocnice Brno Oddeleni Klinicke Onkologie, Brno
  - Masarykuv onkologicky Ustav, Brno
  - Krajska nemocnice Pardubice,oddeleni Radiacni Onkologie, Kyjevska
  - Onkologicka Klinika, Fakultni nemocnice Olomouc, Olomouc
  - Onkologicke Oddeleni, Batova krajska nemocnice Zlin, Zlín
- Hungary (6):
  - National Institute of Oncology, Budapest
  - Szent Imre Korhaz Onkologia, Budapest
  - Szent László Kórház, Onkológia, Budapest
  - Vaszary Kolos Korhaz, Esztergom
  - Petz Aladar County Hospital, Department of Oncology, Győr
  - Baranya megyei Korhaz Onkologial osztaly, Rakoczi
- India (5):
  - Bangalore Institute of Oncology, Bangalore
  - Curie Centre of Oncology, Bangalore
  - Radhakrishan Birla Cancer Centre, Jaipur
  - Jaslok Hospital and Research Centre, Mumbai
  - Sir Ganga Ram Hospital, New Delhi
- Mexico (11):
  - Hospital Clinica del Parque, Chihuahua City, Chihuahua
  - Hospital Universitario "Dr. Angel Leano", Zapopan, Jalisco
  - Hospital y Clinica OCA S.A. De C.V., Monterrey, Nuevo León
  - Hospital Central "Dr. Ignacio Morones Prieto" Departamento de Radioterapia., San Luis Potosí City, San Luis Potosí
  - Hospital regional ISSSTE "Merida", Mérida, Yucatán
  - Centro Estatal de Cancerologia, Chihuahua City
  - Centro Medico ISSEMYM, Metepec
  - Hospital general "5 de Diciembre" ISSSTE, Mexicali
  - Hospital Regional de Especialidades No. 30 IMSS, Mexicali
  - Hospital de Oncologia Centro Medico, Mexico City
  - Instituto Nacional de Ciencias Medicas u Nutricion "Salvador Zubiran", Mexico City
- Romania (5):
  - Fundeni Clinical Institute, Bucharest
  - Trestioreanu Institute of Oncology, Bucharest
  - "I. Chiricuta" Institute of Oncology, Cluj-Napoca
  - Craiova Emergency Clinical County Hospital, Craiova
  - Timisoara City Hospital, Timișoara
- Russia (17):
  - Institute of Medical Radiology, Russian Academy of Medical Science, Obninsk, Kaluga Oblast
  - Cheliabinsk Regional Oncology Center, Chelyabinsk
  - Irkutsk Regional Oncology Center, Irkutsk
  - Clinical Oncology Center, Kazan'
  - Krasnodar City Oncology Center, Krasnodar
  - Blokhin Cancer Research Center, Dept of Clinical Pharmacology and Chemotherapy, Moscow
  - Central Clinical Hospital of the presidentof the Russian Federation, Moscow
  - Hertzen Research Institute of Oncology, Moscow
  - Central Clinical Hospital of the Ministru of Transport n.a. Semashko, Moscow
  - Orenburg, Regional Oncology Center, Orenburg
  - St. Petersburg, Central Research Institute of Radiology, Saint Petersburg
  - Medical Academy of Postgraduate Education, Saint Petersburg
  - Mechnikov State Medical Academy, Saint Petersburg
  - St. Petersburg Oncology Center, Saint Petersburg
  - Samara Oncology Center, Samara
  - Voronezh Regional Clinical Oncology Center, Voronezh
  - Yaroslavl Regional Oncology Center, Yaroslavl
- Ukraine (12):
  - Dnepropetrovsk City Clinical Hospital, Dnipro
  - Donetsk Regional Antitumor Center, Donetsk
  - State Communal Healthcare Institution: Kharkov Regional Clinical Oncological Center, Kharkiv
  - Institute of Oncology under the Academy of Medical Sciences of Ukraine, Kiev
  - Kiev Municipal Clinical Hospital #10, Kiev Center for Biliary, Biliary tracts and Pancreas Surgery, Kiev
  - Krivoy Rog City Oncology Center, Kryvyi Rih
  - Lugansk Regional Clinical Oncological Center, Luhansk
  - Nikolaev Regional Oncology Centre, Mykolayiv
  - Odessa Regional Clinical Hospital, Odesa
  - Vinnitsa Regional Clinical Oncology Center, Vinnitsa
  - Zaporozhye Medical Academy of Postgraduate Education, Zaporizhzhya
  - Zhitomir Regional Clinical Hospital n.a. O.F. Gerbachevsky, Zhytomyr

REFERENCES:
- See also: Threshold Pharmaceuticals Website — http://www.thresholdpharm.com